CLINICAL TRIAL: NCT05455294
Title: A Phase 1 Study of Triplet Therapy With Navitoclax, Venetoclax, and Decitabine for High-risk Myeloid Malignancies
Brief Title: Combination Navitoclax, Venetoclax and Decitabine for Advanced Myeloid Neoplasms
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jacqueline Garcia, MD (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor-Investigator, Jacqueline Garcia, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-263
Record Dates: First submitted 2022-07-05; First posted 2022-07-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Myeloid Malignancy; Myelodysplastic Syndromes; Myelofibrosis; Acute Myeloid Leukemia; Myeloproliferative Neoplasm
Keywords: Myeloid Malignancy; Myelodysplastic Syndromes; Myelofibrosis; Acute Myeloid Leukemia; Myeloproliferative Neoplasm; MDS-myeloproliferative neoplasm
MeSH Terms: conditions — Myelodysplastic Syndromes; Primary Myelofibrosis; Leukemia, Myeloid, Acute; Myeloproliferative Disorders | interventions — navitoclax; venetoclax; Decitabine

STUDY DESIGN:
Intervention Model Description: This is a Phase 1 study with a dose escalation design and an expansion cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Level 0: Decitabine + Venetoclax + Navitoclax [AML and Non-AML] (Experimental): Dose Level 0 [AML and Non-AML]
  Decitabine [intravenously (IV) preferred]
  Venetoclax Cycle 1: ramp-up days 1-2 and days 3-14 absence of strong/moderate CYP3A inhibitor and reduced doses dependent on presence of moderate or strong CYP3A inhibitor Cycle 2+: dosing days 1-14
  Navitoclax Cycle 1: dosing days 3-14; Cycle 2+: dosing on days 1-14
  Cycle length=28 days Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: Navitoclax; Drug: Venetoclax; Drug: Decitabine
- Dose Level 1: Venetoclax + Decitabine + Navitoclax [AML and Non-AML] (Experimental): Dose Level 1 [AML and Non-AML]
  Decitabine [intravenously (IV) preferred] Cycle 1+: dosing on days 1-5
  Venetoclax [orally] Cycle 1: ramp-up starting on day 1-2 then days 3-14 continued dosing in absence of strong/moderate CYP3A inhibitor and reduced doses dependent on presence of moderate or strong CYP3A inhibitor Cycle 2+: dosing days 1-14
  Navitoclax [orally] Cycle 1: Dosing days 3-14 Cycle 2+: dosing on days 1-14
  Cycle length=28 days Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: Navitoclax; Drug: Venetoclax; Drug: Decitabine
- Dose Level 2: Venetoclax + Decitabine + Navitoclax [AML] (Experimental): Dose Level 2 [AML]
  Decitabine [intravenously (IV) preferred] Cycle 1+: dosing on days 1-5
  Venetoclax [orally] Cycle 1: ramp-up on day 1-2, days 3-21 continued dosing in absence of strong/moderate CYP3A inhibitor and reduced doses dependent on presence of moderate or strong CYP3A inhibitor Cycle 2+: dosing on days 1-21
  Navitoclax [orally] Cycle 1: dosing on days 3-14 Cycle 2+: dosing on days 1-14
  Cycle length=28 days Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: Navitoclax; Drug: Venetoclax; Drug: Decitabine
- Dose Level -1: Venetoclax + Decitabine + Navitoclax [Non-AML] (Experimental): Dose Level -1 [Non-AML]
  Decitabine [intravenously (IV) preferred] Cycle 1+:dosing [intravenously (IV) preferred] on days 1-3
  Venetoclax [orally] Cycle 1: ramp-up of starting day 1-2 then days 3-7 continued dosing in absence of strong/moderate CYP3A inhibitor and reduced doses dependent on presence of moderate or strong CYP3A inhibitor Cycle 2+: dosing on days 1-7
  Navitoclax [orally] Cycle 1: Dosing days 3-14 Cycle 2+: continued dosing on days 1-14
  Cycle length=28 days Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: Navitoclax; Drug: Venetoclax; Drug: Decitabine
- Recommended Phase 2 Dose Level: Venetoclax + Decitabine + Navitoclax [AML and Non-AML] (Experimental): RP2D [AML and Non-AML]
  Decitabine [intravenously (IV) preferred] To be determined based on dose escalation design.
  Venetoclax [orally] To be determined based on dose escalation design.
  Navitoclax [orally] To be determined based on dose escalation design.
  Cycle length=28 days Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: Navitoclax; Drug: Venetoclax; Drug: Decitabine

INTERVENTIONS:
Drug: Navitoclax — See Arm Description
  Other Names: ABT-263
Drug: Venetoclax — See Arm Description
  Other Names: Venclexta
Drug: Decitabine — See Arm Description
  Other Names: Dacogen

SUMMARY:
The purpose of this research study is to test the safety of a new three drug combination of navitoclax, decitabine, and venetoclax to treat advanced myeloid malignancies.

The names of the drugs involved in this study are:

* Venetoclax
* Decitabine
* Navitoclax

DETAILED DESCRIPTION:
This is a phase 1 study to determine the safety, dosing schedule and recommended phase 2 dose of a triplet therapy with navitoclax, venetoclax, and decitabine for patients with the four high-risk myeloid malignancy subgroups of acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), myeloproliferative neoplasm (MDS/MPN) and myelofibrosis accelerated phase (MF-AP).

The U.S. Food and Drug Administration (FDA) has not approved the combination of venetoclax, navitoclax, and decitabine navitoclax as a treatment for any disease.The FDA has approved the combination of venetoclax and decitabine for acute myeloid leukemia (AML) and decitabine given alone is approved for myelodysplastic syndrome (MDS).

The research study procedures include screening for eligibility, study treatments, and blood tests and bone marrow biopsies to assess response to treatment.

Participants will receive the study treatment regimen as long as it is effective.

It is expected that about 36 people will take part in this research study.

AbbVie, a pharmaceutical company, is supporting this research study by providing funding and the study drugs navitoclax and venetoclax.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Subjects must have a diagnosis of one of the following:

  * Myelofibrosis in accelerated phase (AP-MF), defined by WHO as 10-19% blasts in either bone marrow or blood. There is no requirement for prior therapy.
  * Myelofibrosis in blast phase (BP-MF), defined as ≥ 20% blasts in either bone marrow or blood. There is no requirement for prior therapy.
  * Untreated secondary AML (s-AML), which includes subjects with therapy-related disease or known antecedent MDS or MDS/MPN. All these subjects must be ineligible or not recommended for any available approved therapy as determined by the treating provider. For subjects with known antecedent MDS or MDS/MPN, they must have received prior HMA therapy (minimum number of cycles are not required in this setting).
  * MDS/MPN overlap syndromes (e.g. CMML) with ≥ 5% blasts in either bone marrow or blood. No requirements for prior therapy.
  * MDS with excess blasts defined as ≥ 5% blasts in either bone marrow or blood must be ineligible for any available approved therapy including intensive chemotherapy and immediate allogeneic stem cell transplant per treating investigator and must meet at least one of the following criteria: 1) persistent disease despite prior exposure to venetoclax plus HMA for at least 3 cycles, 2) disease progression per IWG 2006 criteria on venetoclax plus HMA or on M15-954 protocol, or 3) persistent disease after at least four cycles of any HMA-based therapy.
* ECOG performance status ≤ 2 (see Appendix A)
* Baseline platelet count ≥ 25 x 109/L
* Subjects must have adequate organ function as defined below:

  * Aspartate transaminase (AST) and alanine transaminase (ALT) < 3 x ULN
  * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
  * Subject must have adequate renal function as demonstrated by a creatinine clearance ≥ 45 mL/min; calculated by the Cockcroft Gault formula
  * aPTT ≤ 1.5 x ULN
  * INR ≤ 1.5 x ULN
* Prior treatment-related toxicities must be grade 1 or baseline except for alopecia.
* Moderate/strong inhibitors of CYP3A are allowed if they cannot be substituted; however, patients must be on these agents for at least 2-3 days prior to treatment start. (See section 5.5 for details on concomitant medications and dose adjustment.)
* If female, subject must be either :

  * Postmenopausal (surgically sterile or age > 55 years with no menses for 12 or more months without an alternative medical cause or age greater than or equal to 55 or less with no menses for 12 or more months without an alternative medical cause and an FSH level > 40 IU/L); or
  * Of children bearing potential. These subjects must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Subject must agree to have a negative urine or serum beta-HCG test result during screening and repeated within 7 days prior to study drug (local labs are allowed) to be eligible.
* Subject must voluntarily sign and date an informed consent
* Subjects must be able to swallow pills

Exclusion Criteria:

* Subject cannot have had prior navitoclax or any BCL-XL therapy. Otherwise, there are no restrictions on any other prior therapies. Prior venetoclax is allowed.
* Subject is eligible and willing to receive intensive chemotherapy for their specific disease.
* Anti-leukemic therapy within 14 days of first day of study treatment except for hydroxyurea. If on hydroxyurea, then subject needs to be off hydroxyurea at least 3 days prior to first dose of study treatment. If on venetoclax, then a wash-out period of at least five times the half-life of the treatment.
* Subject with known and active concurrent malignancy requiring treatment. Subjects with basal or squamous skin cancers or carcinomas in situ are allowed. Exception: hormonal or topical therapies are allowed.
* Subject has known active/uncontrolled HIV and on contraindicated medication due to drug-drug CYP inducer interaction. HIV testing is not required.
* Subject has known and active CNS involvement with AML.
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * Uncontrolled and/or active systemic infection (viral, bacterial or fungal). Controlled infections are allowed.
  * Chronic, active hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate. Subjects that have prior HCV that has been definitively treated with negative HCV viral load prior to study initiation and no evidence of cirrhosis are allowed to participate.
* Recent diagnosis of myocardial infarction or worse heart failure within the last six months.
* Treatment with any moderate or strong CYP3A inducers (see Appendix D for examples) within 7 days prior to the first dose of study drug.
* Administration or consumption of any of the following within 3 days prior to the first dose of study drug:

  * Grapefruit or grapefruit products
  * Seville oranges (including marmalade containing Seville oranges)
  * Star fruit
* White blood cell count (WBC) greater than or equal to 25 x 109/L. Exception: Subjects with myelofibrosis or MDS/MPN overlap syndrome may enter study with WBC greater than or equal 25 x 109/L on the first day of therapy only if the absolute blast count is < 5 x 109/L; hospitalization for subjects with this particular disease subset is required during dose ramp-up of venetoclax for TLS monitoring. This criterion is intended to exclude AML patients at high risk of TLS, but permit entry of patients with MF or CMML who frequently have leukocytosis without AML transformation who are at low risk for TLS.
* Ongoing requirement for anticoagulation with the exception of low-dose anticoagulation medications used to maintain patency of a central venous catheter or for deep venous thrombosis prophylaxis. Antiplatelet agents such as aspirin and clopidogrel are not allowed if platelet count < 50 x 109/L.
* Known history of immune thrombocytopenia that previously required therapy.
* Known history of platelet refractoriness and HLA alloimmunization prior to study start.
* History of serious or life-threatening bleeding in last 12 months that has not been definitively treated.
* Uncontrolled, systemic infection (viral, bacterial, or fungal). Antibiotic use is permitted. (See Section 5.5 for concomitant drugs)
* Active and known SARS-CoV-2 infection.

  * If a subject has signs/symptoms suggestive of SARS-CoV-2 infection, then the subject must undergo molecular (e.g. PCR) testing to rule out SARS-CoV-2 infection.
  * Subjects positive for active SARS-CoV-2 infection may re-screen after they meet either criteria A or B indicating SARS-CoV-2 infection has resolved with viral clearance: A) ≥14 days since first the PCR test result in an asymptomatic subject; OR B) ≥14 days since recovery, defined as resolution of fever without use of anti-pyretics and improvement in symptoms.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the subject inappropriate for enrollment into this study.
* Vaccination with live, attenuated vaccines ≤4 weeks prior to initiation of study treatment or anticipation of need for such a vaccine during the study. All other recommended vaccinations including COVID19 is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | The observation period for RP2D evaluation was the first 28 days (cycle 1) of treatment.
  The RP2D is the minimally safe and biologically effective dose. The minimally safe dose is the highest dose level at which <2 of 6 participants experience a dose limiting toxicity (DLT). See subsequent primary outcome for the DLT definition. With respect to safety, the RP2D will also consider laboratory evidence of platelet recovery. Evaluation of efficacy will be done in real time prioritizing full complete response (see subsequent secondary outcome for the objective response criteria) when possible for AML/MDS/MDS-MPN and transfusion independence/blast reduction/TSS improvement/splenic reduction for myelofibrosis.
Dose Limiting Toxicity (DLT) | The observation period for DLT evaluation was the first 28 days (cycle 1) of treatment.
  DLT is defined by hematologic or non-hematologic adverse event (AE) per protocol (section 5.4); A treatment-related death is a DLT; AEs are graded based on NCI CTCAE v5.0 and must be considered unrelated to the underlying disease or co-morbidity to be a DLT.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Bone marrow evaluation for disease response is performed end of C1, C2, every 2 cycles until CR/CRi and then every 3 cycles. Each cycle is 28 days. Time frame is indefinite as based on maximum treatment duration which is not fixed.
  Response criteria follows consensus guidelines set forth by international working groups for MF, MDS (MDS: CR, marrow CR, PR, HI), MDS/MPN overlap syndromes, and AML. ORR, evaluated by disease type, is defined as the proportion of participants achieving objective response per protocol (section 11.1) on treatment:
  * AP/BP-MF: CR, PR, Clinical Improvement
  * MDS: CR, marrow CR, PR, HI
  * CMML: CR, PR, marrow CR
  * s-AML: CR, CRi, CRp
Median Progression-Free Survival (PFS) | Bone marrow evaluation for disease response is performed days 22-28 of C1, end of C2, every 2 cycles (cycle end) until CR/CRi and then every 3 cycles. Off treatment, disease is assessed every 4 months up to 2 years.
  Progression-free survival based on the Kaplan-Meier method is defined as the time from study treatment to evidence of progression (for MDS per IWG 2006 criteria; for AML per ELN 2017 criteria; for MF per IWG criteria, defined per protocol section 11.1) or at death due to any cause including underlying disease. Participants alive without disease progression are censored at date of last follow up.
Overall Survival (OS) | Survival is assessed in long-term follow-up every 4 months up to 2 years.
  OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.

OTHER OUTCOMES:
Navitoclax Target Dose Rate | While on study treatment for up 1 year
  The navitoclax target dose rate is the proportion of participants without navitoclax dose modifications on treatment per protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline S Garcia, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu